CLINICAL TRIAL: NCT00757328
Title: EPIDEP. Epidemiologic Study in Bipolar Depression: Evaluation of the Usual Clinical Practice of Psychiatrists in Spain
Brief Title: Treatment Clinical Practice in Bipolar Depression in Spain
Acronym: EPIDEP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, PhD, Local MC Neuroscience Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2008/3
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression Treatment
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Ambulatory bipolar I and II patients, clinically stabilized for at least the two months prior to recruitment and who had at least one acute episode (depressive, manic, hypomanic or mixed) within the year prior to recruitment.

SUMMARY:
Cross-sectional observational, non interventional, multicenter study of retrospective review of clinical records of ambulatory followed up bipolar patients in order to record epidemiological aspects of the course of the disorder, more specifically of bipolar depression episodes and the clinical practices carried out by psychiatrists in Spain in bipolar depressive episodes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of Bipolar Disorder I or II (DSM-IV-TR) in ambulatory follow-up
* Evolution of the bipolar diagnoses inferior to 10 years
* Having recorded in the patient's clinical history the clinical management of at least two bipolar depressive episodes

Exclusion Criteria:

* Not having enough information recorded in the clinical history for the essential measurement variables
* To have taken part in other study in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult bipolar I or II patients with no more than 10 years of evolution of the bipolar disorder, with continued assistance in ambulatory settings and whose psychiatrist has recorded the treatment strategy used for of at least 2 depressive episodes within the patients' bipolar condition in the clinical history
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2008-07; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacological treatments used in Spain by Psychiatrists in the management of bipolar depressive episodes in first and second line | Last two bipolar episodes recorded in tha patient's clinical history

SECONDARY OUTCOMES:
Non pharmacological treatments used in Spain by Psychiatrists in the management of bipolar depressive episodes in first and second line | Last two bipolar episodes recorded in tha patient's clinical history
Description of the course of the patients' bipolar disorder | Course of the disorder recorded in the patient's clinical history

CONTACTS AND LOCATIONS:
Locations (23):
- Spain (23):
  - Research Site, Santander, Cantabria
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Santiago C., La Coruna
  - Research Site, Palma M, Mallorca
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Bilbao, Vizcaya
  - Research Site, Alicante
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Huesca
  - Research Site, Las Palmas
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid